CLINICAL TRIAL: NCT00761072
Title: An Evaluation of RemifentanilPropofol Infusion in Pediatric Spinal Surgery
Brief Title: Remifentanil Propofol Infusion in Pediatric Spinal Surgery
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-05-6048
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Spinal Fusion
Keywords: Propofol; Remifentanil; Total Intravenous Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: The source of data will be from spinal surgery procedures performed at CHOP from 4/1/07 to 3/31/08 using a TIVA anesthetic technique of propofol/remifentanil infusions

SUMMARY:
Total intravenous anesthesia(TIVA) is a commonly used anesthetic technique. Although TIVA can be accomplished with a variety of drug combinations, infusions of Propofol and Remifentanil are often used with dosage adjusted manually by the anesthesia provider.The pharmacokinetics of these drugs are well understood, and that knowledge has led to the development of computer controlled infusion pumps that can administer the drugs based upon pharmacokinetic models. Computer controlled infusion schemes automatically adjust the drug administration based upon pharmacokinetic models which typically dictate a tapering infusion scheme. When one considers the dosage of a computer controlled infusion it is obvious that manually imitating a similar scheme may be difficult.This study will evaluate manually controlled infusion schemes using the models built into the Applied Medical Visualizations (Medvis) display and compare the manual dosage schemes to the predicted effect site concentrations and pharmacodynamic effect.

DETAILED DESCRIPTION:
During Total intravenous anesthesia (TIVA), the anesthetic propofol and the opioid remifentanil are often used together. Previous studies have demonstrated the synergy between these combinations of medications. From these data, drug interaction models have been developed to pair drug effect-site concentrations with event markers of interest to the clinical anesthesiologist. For example, the amount of remifentanil and propofol typically required during the induction of anesthesia to cause loss of responsiveness to verbal or moderate stimuli has been studied. Likewise, the blood concentration levels present during emergence from anesthesia have been explored describing levels typically present for patients to return to consciousness.

The purpose of this study is to retrospectively analyze the infusion doses of both remifentanil and propofol for pediatric patients undergoing spinal fusion surgery at CHOP. These data will be applied to the pharmacokinetic models to determine the predicted effect site concentration, and the relationship of that concentration to the 50% and 95% doses as predicted by the model.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female patients age 0 to 18 years old
2. Spinal surgery at CHOP between 4/1/07 and 3/31/08
3. Complete CompuRecord Anesthesia documentation
4. Use of Propofol and Remifentanil infusions as primary anesthetic technique

Exclusion Criteria:

1. Chronic opioid or benzodiazepine medication use prior to surgery
2. Use of other anesthetic infusions (i.e. Ketamine/Fentanyl) during TIVA
3. Use of Neuraxial opioids
4. Use of other Induction medications (i.e. Sodium Thiopental)

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients having spinal surgery procedures completed at CHOP from April 2007 through March 2008
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary purpose of the study is to investigate the consistency in predicted effect site concentrations that result from manual administration of propofol and remifentanil for TIVA | Between 4/1/2007 until 3/31/2008.

SECONDARY OUTCOMES:
The secondary objectives are to determine the variability in propofol-remifentanil TIVA dosing in a population of surgical patients | 4/1/2007 to 3/39/2008
The secondary objectives are to determine the variability in propofol-remifentanil TIVA dosing in a population of surgical patients | 4/1/2007 - 3/31/2008
To gain insight into the potential benefit of using a real time display of predicted serum levels and pharmacodynamic response to guide manual drug infusion for TIVA | 4/1/2007 - 3/31/2009

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Feldman, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States